CLINICAL TRIAL: NCT04668846
Title: A Multicenter Sample Collection Study Utilizing DermTech's Non-invasive Adhesive Patch Biopsy Kits in Subjects With a Variety of Dermatologic Conditions
Brief Title: A Sample Collection Study Utilizing DermTech's Non-invasive Adhesive Patch Biopsy Kits
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DermTech (Other)
Responsible Party: Sponsor
Other Study IDs: 17-06
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-03

CONDITIONS: Dermatologic Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non-invasive collected skin samples will be collected and banked for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-invasive sample collection of skin tissue — Both lesional and non-lesional skin will be sampled with up to 24 adhesive patches.

SUMMARY:
This sample collection study will recruit subjects with a variety of skin conditions from up to 15 geographically dispersed sites in the United States. Skin samples will be collected with the DermTech Adhesive Patch Kit from both lesional and non-lesional skin. Subjects may also be asked to return at a future data for additional collections. Collected skin samples will be analyzed for gene expression information, DNA and the microbiome.

DETAILED DESCRIPTION:
This is a multi-center, sample collection study to obtain skin tissue for gene expression, DNA mutation, microbiome and related analyses from subjects with dermatologic conditions. After subjects are consented for the study, site staff will collect skin tissue from the subject using DermTech's non-invasive skin collection kit. Skin samples will be collected from both lesional and non-lesional skin as applicable.

Additional skin tissue may be collected from the lesion and non-lesional area with the DermTech non-invasive skin collection kit at a later time point as directed by DermTech to track the dermatologic condition for progression, improvements or lack of response to standard of care therapy.

Each Dermtech non-invasive skin collection kit will consist of the sequential application of up to 24 individual patches to lesional and non-lesional areas. Sites should apply the DermTech patches to the most severe lesion(s).

Dermatologic conditions include but are not limited too; atopic dermatitis, atopic asthma, skin cancers (i.e., basal, and squamous carcinoma, melanoma, etc.), lupus, rheumatoid and psoriatic arthritis, gutate and plaque psoriasis, palmoplantar psoriasis, palmoplantar contact dermatitis, fungal infections and cutaneous T cell Lymphoma. Skin tissue will be collected using DermTech's proprietary adhesive patch skin biopsy kit and extracted for analysis at DermTech's CLIA and CAP Laboratory. Analysis of the samples will include gene expression signatures and DNA mutation as well as microbiome analyses associated with the medical conditions of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 21 years of age;
2. Have a dermatologic condition of interesting including but not limited too; atopic dermatitis, atopic asthma, skin cancers (i.e., basal, and squamous carcinoma, melanoma, etc.), lupus, rheumatoid and psoriatic arthritis, gutate and plaque psoriasis, palmoplantar psoriasis, palmoplantar contact dermatitis, fungal infections and cutaneous T cell Lymphoma that can be non-invasively biopsied with DermTech's adhesive patch kit;
3. Willing to allow additional DermTech adhesive patch biopsies to be performed; and
4. Willing to provide informed consent to participate in this trial.

Exclusion Criteria:

1. Required a surgical biopsy or excision prior to a PLA on that lesion of interest;
2. Has an ulcerated or bleeding lesion that could cofound the PLA results;
3. Has a suspicious lesion(s) in an area that was previously surgically biopsied;
4. Has an allergy to tape or latex rubber; and
5. Receipt of any investigational drug therapy within four weeks of study enrollment, or concurrent participation in another interventional clinical study deemed by the treating physician to potentially influence this study.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with a variety of dermatologic conditions will have both lesional and non-lesional skin collected using the DermTech non-invasive adhesive patch kit. Dermatologic conditions include but are not limited too; atopic dermatitis, atopic asthma, skin cancers (i.e., basal, and squamous carcinoma, melanoma, etc.), lupus, rheumatoid and psoriatic arthritis, gutate and plaque psoriasis, palmoplantar psoriasis, palmoplantar contact dermatitis, fungal infections and cutaneous T cell Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Gene Expression Analysis | 24 months
  To collect skin tissue from subjects with a variety of dermatologic conditions, both lesional and non-lesional areas to analyze for unique gene signatures

CONTACTS AND LOCATIONS:
Overall Officials: James Rock, MS, Study Director — DermTech
Locations (2):
- United States (2):
  - Elizabeth S. Robinson, MD, Denver, Colorado
  - Skin Care Research, LLC, Boca Raton, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yao Z, Moy R, Allen T, Jansen B. An Adhesive Patch-Based Skin Biopsy Device for Molecular Diagnostics and Skin Microbiome Studies. J Drugs Dermatol. 2017 Oct 1;16(10):979-986. PMID 29036251
- [Background] Krueger G, Jansen B, Yao Z. Non-Invasive Gene Expression Analysis Assay for Psoriasis. Poster Presentation American Academy of Dermatology. March 2017.